CLINICAL TRIAL: NCT00734721
Title: Fear of Intravitreal Injection - Assessment of Psychological Strain and Potential Contributing Factors
Brief Title: Assessment of Psychological Strain and Perioperative Fear in Intravitreal Injections
Acronym: FIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Ziemssen/Dr, University Eye Hospital Tuebingen
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: UEH-2007FIV
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2008-08

CONDITIONS: Age-related Macular Degeneration; Stress
Keywords: intravitreal injection
MeSH Terms: conditions — Macular Degeneration | interventions — Perioperative Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): Presentation of factual information video
  Interventions: Behavioral: Preoperative information and perioperative care
- B (Active Comparator): Presentation of injection syringe/needle
  Interventions: Behavioral: Preoperative information and perioperative care
- C (Active Comparator): Presentation of emotional information video
  Interventions: Behavioral: Preoperative information and perioperative care
- D (Active Comparator): Stress relaxation music
  Interventions: Behavioral: Preoperative information and perioperative care

INTERVENTIONS:
Behavioral: Preoperative information and perioperative care — Patients receive different information and care in addition to the basic medical consultation.

SUMMARY:
1. Intravitreal injection can induce perioperative stress for the patients.
2. Different factors can modulate the pre-operative fear and physiologic reaction.

DETAILED DESCRIPTION:
The aim of the study is to assess the influence of perioperative factors on objective outcome measures, which indicate the physiologic stress reaction.

ELIGIBILITY:
Inclusion Criteria:

* First intravitreal injection received ever

Exclusion Criteria:

* No known affective or mental disorder
* Condition does not allow standardized survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Objective parameters of stress reaction | 12 months

SECONDARY OUTCOMES:
Subjective Response (state-trate anxiety) in respect of coping behaviour | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Tübingen, Baden-Wurttemberg, Germany